CLINICAL TRIAL: NCT00121212
Title: Positron Emission Tomography in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000434994; R01CA101734 (NIH); P30CA091842 (NIH); WU-03-0315
Record Dates: First submitted 2005-07-19; First posted 2005-07-21 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Surgery - Negative PET scan (Active Comparator): If patient is candidate for surgery with curative intent or staging lymphadenectomy, he will be enrolled in the study. If patient's PET scan is negative, the patient will receive the curative therapy and be followed for recurrence.
  Interventions: Procedure: carbon-11 acetate PET scan
- Surgery - Positive PET scan (Experimental): If patient is candidate for surgery with curative intent or staging lymphadenectomy, he will be enrolled in the study. If patient's PET scan is positive, the patient will receive the curative therapy and be followed for recurrence or receive alternative therapy.
  Interventions: Procedure: carbon-11 acetate PET scan
- Radiation therapy Negative or Positive PET scan (Active Comparator): If patient is candidate for radiation therapy with curative intent, he will be enrolled. If PET scan is negative he will receive curative therapy and be followed for PSA recurrence. If PET scan is positive he may receive confirmatory studies and then if negative, not indicated, or refused he will receive curative therapy be followed for PSA recurrence. If PET scan is positive and received positive confirmatory studies he will receive curative therapy and followed for recurrence.
  Interventions: Procedure: carbon-11 acetate PET scan

INTERVENTIONS:
Procedure: carbon-11 acetate PET scan

SUMMARY:
RATIONALE: Diagnostic procedures, such as positron emission tomography using carbon-11 acetate, may help find metastases from prostate cancer and may help predict whether prostate cancer will come back after treatment.

PURPOSE: This clinical trial is studying how well positron emission tomography using carbon-11 acetate works in finding metastases and predicting recurrence in patients with prostate cancer who are at risk for recurrence after treatment.

DETAILED DESCRIPTION:
The overall goal of this project is determination of the role of PET in patients with newly diagnosed medium- and high-risk prostate cancer in whom the standard clinical and imaging workup is negative. Thus, the incremental value of PET will be determined in this important group.

ELIGIBILITY:
Inclusion Criteria

* Newly diagnosed prostate cancer
* Has completed conventional staging examinations, including biopsy with Gleason score, CT scan of the abdomen and pelvis, and whole-body bone scintigraphy AND conventional staging examinations negative
* Candidate for curative radical prostatectomy OR curative radiotherapy OR staging lymphadenectomy prior to surgery
* Deemed to be at medium or high risk for recurrence after initial curative treatment, as defined by 1 of the following criteria:

  * Gleason score 7 AND prostate-specific antigen (PSA) 10-20 ng/mL
  * Gleason score ≥ 8 AND PSA < 10 ng/mL
  * Gleason score ≥ 8 AND PSA > 10 ng/mL
  * Any Gleason score AND PSA > 20 ng/mL

Exclusion Therapy:

* Not a candidate for treatment by surgery or radiation therapy with curative intent
* Inability to give informed consent
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of other cancer present within the last 5 years

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2003-07; Primary Completion 2010-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Determine the role of AC-PET in changing initial patient management | Completion of patient treatment

SECONDARY OUTCOMES:
Determine the value of AC-PET in predicting recurrence | Minimum of 2 years and maximum of 5 years
Assess the performance of AC-PET for detection of lymph node metastasis by comparison with biopsy. | Minimum of 2 years and maximum of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Farrokh Dehdashti, MD, Study Chair — Washington University Siteman Cancer Center
Locations (1):
- Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri, United States